CLINICAL TRIAL: NCT05903209
Title: A Study to Evaluate Accuracy and Validity of Chang Gung Pneumothorax Detection Software Compared With Reference by Qualified Physicians
Brief Title: A Study to Evaluate Chang Gung Pneumothorax Detection Software
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200871B0
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-05

CONDITIONS: Pneumothorax
Keywords: artificial intelligence
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Software diagnosis: Software diagnosis with gold standard of 3 doctors' interpretation.
  Interventions: Device: Chang Gung Pneumothorax Detection Software

INTERVENTIONS:
Device: Chang Gung Pneumothorax Detection Software — The Chang Gung Pneumothorax Detection Software is an independent software as a medical device, which inputs digital Chest X-Ray to automatically detect whether there is a pneumothorax. The inferred results output by this software can assist clinicians or professional medical personnel to identify whether a patient has pneumothorax.
  This product is only used to analyze the digitized Chest X-Ray DICOM of patients over 20 years old and under 100 years old.

SUMMARY:
The Chang Gung Pneumothorax Detection Software is a medical software that can automatically detect whether there is a pneumothorax in Chest X-Ray. The purpose of this study is to verify whether the Chang Gung Pneumothorax Detection Software can correctly identify patients with pneumothorax in Chest X-Ray. The results of the software analysis will be used for the performance of the software on the primary and secondary outcomes.

DETAILED DESCRIPTION:
This clinical trial is a retrospective study. DICOM images of de-identified Chest X-Ray were collected from 6 hospitals of Chang Gung Memorial Hospital from January 1, 2006 to December 31, 2020. The test set of 5,347 items was established, and total of 344 cases will be sampled by simple random stratification, including 172 cases with pneumothorax and 172 cases without pneumothorax. The image must be in DICOM format.

Follow-up by three specialist physicians to interpret the presence or absence of pneumothorax, the result will be the standard of this test (Reference). After confirming the correct standard of each Chest X-Ray, the Chest X-Ray will be put into Chang Gung Pneumothorax Detection Software, and analyzed by the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The case were over 20 years old and under 100 years old.
* DICOM format.
* Brand model of Canon.
* DICOM resolution length range (700-3400 pixels), width range (490-3600 pixels).
* poster-anterior view(PA-view) of chest X-ray

Exclusion Criteria:

* The chest X-ray contains items that affect interpretation, such as chest tubes, endotracheal tubes, and heart rhythm regulators, but does not include patches and circuits used in electrocardiograms.
* The chest X-ray that are difficult to interpret due to poor image quality.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study, and the data comes from the Chang Gung Medical Research Database(CGRD) which was an database form 6 hospitals of Chang Gung Memorial hospital. According to inclusion and exclusion criteria, Chest X-ray data from the database during 2006.01.01~2020.12.31 was collected.
Sampling Method: Probability Sample
Enrollment: 344 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | baseline
  The rate of test results that correctly indicate the presence.

SECONDARY OUTCOMES:
Specificity | baseline
  The rate of test results that correctly indicate the absence.
Area Under the receiver operating characteristic Curve | baseline
  A graphical plot that illustrates the diagnostic ability of a binary classifier system as its discrimination threshold is varied.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Fu Kuo, Study Chair — Associate Professor and Director Division of Rheumatology
Locations (1):
- Chang Gung memorial hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebrahimi A, Yousefifard M, Mohammad Kazemi H, Rasouli HR, Asady H, Moghadas Jafari A, Hosseini M. Diagnostic Accuracy of Chest Ultrasonography versus Chest Radiography for Identification of Pneumothorax: A Systematic Review and Meta-Analysis. Tanaffos. 2014;13(4):29-40. PMID 25852759
- [Background] Nagarsheth K, Kurek S. Ultrasound detection of pneumothorax compared with chest X-ray and computed tomography scan. Am Surg. 2011 Apr;77(4):480-4. PMID 21679560
- [Background] Nandipati KC, Allamaneni S, Kakarla R, Wong A, Richards N, Satterfield J, Turner JW, Sung KJ. Extended focused assessment with sonography for trauma (EFAST) in the diagnosis of pneumothorax: experience at a community based level I trauma center. Injury. 2011 May;42(5):511-4. doi: 10.1016/j.injury.2010.01.105. Epub 2010 Feb 10. PMID 20149371
- [Background] Lachin JM. Properties of simple randomization in clinical trials. Control Clin Trials. 1988 Dec;9(4):312-26. doi: 10.1016/0197-2456(88)90046-3. PMID 3203523
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415